SCB01A for Metastatic Squamous Cell Head and Neck Cancer

# Statistical Analysis Plan: Mock-up Tables and Figures

Version 3.0, 14DEC2018

**Protocol Number: SCB01A-22** 

An Open-Label, Phase II Study to Evaluate the Efficacy and Safety of SCB01A in Subjects with Recurrent or Metastatic Squamous Cell Head and Neck Cancer Who Have Failed Platinum-Based Treatment

Protocol version: 1.0/19-Dec-2016 Sponsor: SynCore Biotechnology Co., Ltd.



# **Statistical Analysis Plan:** Mock-up Tables and Figures SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### **Table of Contents**

| St | atistical Ana | ılysis Plan: Mock-up Tables and Figures | 1 |
|---|---|---|---|
| Ta | ble of Cont | ents | 2 |
| 1 | Statistic | al Changes from Study Protocol | 3 |
| | 1.1 PK | Analysis | |
| | | jective response rate (ORR) Definition | |
| 2 | Mock-uj | p Tables and Figures | 3 |
| 3 | Change | From Preceding Version of Statistical Analysis Plan | 5 |
| | 3.1 SA | P 2.0: Progression Free Survival (PFS) Estimation | 5 |
| | 3.2 SA | P 3.0: Response Evaluation | 6 |
| 14 | TABLES | S and FIGURES | 7 |
| | 14.1 DE | EMOGRAPHIC DATA AND BASELINE CHARACTERISTICS | 7 |
| | 14.1.1 | Screen Failures and Subject Disposition by Study Site | |
| | 14.1.2 | Study Visits, Study Termination, Subject Disposition and Protocol Deviation | |
| | 14.1.3 | Demographic Data, Smoking Status and Betelnut Consumption | |
| | 14.1.4 | Head and Neck Squamous Cell Carcinoma History & Tumor Staging | |
| | 14.1.5 | General Medical History | |
| | 14.1.6 | Study Drug Administration | |
| | 14.2 EF | FICACY DATA | |
| | 14.2.1 | Objective Response Rate | |
| | | • | |
| | | FETY DATA | |
| | 14.3.1 | Treatment Emergent Adverse Events – Subject Based Analyses | |
| | 14.3.2 | Clinical Relevance of Laboratory Assessment – Hematology | |
| | 14.3.3 | Clinical Relevance of Laboratory Assessment – Biochemistry | |
| | 14.3.4 | Clinical Relevance of Laboratory Assessment – Coagulation | |
| | 14.3.5 | Clinical Relevance of Laboratory Assessment – Urinalysis | |
| | 14.3.6 | Toxicity Grade of Laboratory Assessment – Hematology | |
| | 14.3.7 | Toxicity Grade of Laboratory Assessment – Biochemistry | |
| | 14.3.8 | Toxicity Grade of Laboratory Assessment – Coagulation | |
| | 14.3.9<br>14.3.10 | Toxicity Grade of Laboratory Assessment –Urinalysis | |
| | 14.3.10 | Nerve Conduction Velocity Examination | |
| | 14.3.11 | Electrocardiogram (ECG, EKG) | |
| | 14.3.12 | Physical Examination | |
| | 17.5.15 | THYSICAL DAMINIANUIL | ∠∪ |

# 

# Statistical Analysis Plan: Mock-up Tables and Figures

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### 1 Statistical Changes from Study Protocol

The statistical analysis methods will follow study protocol version 1.0, 19DEC2016, exceptions and clarifications are described below:

#### 1.1 PK Analysis

Pharmocokinetics Sampling will be bio-analyzed, and PK Parameters will be calculated by Protech Pharmaservices Corporation. All PK and PK parameter data will be provided to sponsor directly, no data handling, data listing nor statistical analysis on such data will be done by A2 Healthcare.

#### 8.6. PK Analysis

The blood samples will be assayed for SCB01A and PK parameters (maximum plasma concentration [Cmax], clearance [CL], volume of distribution [Vd], half-life [t1/2], elimination constant [Kel], mean residence time [MRT] and time to maximum concentration [Tmax]) will be determined and presented graphically and descriptively (as appropriate).

#### 1.2 Objective response rate (ORR) Definition

ORR is defined as the percentage of subjects who have achieved confirmed CR and PR during treatment phase, according to RECIST v1.1. Not-confirmed CR or PR, or withdraw for DLT are counted as non-responder. There are 5 subjects who are not evaluated due to clinical disease progression or AE/SAE. Tumor non-evaluable subjects are tend to be treatment failure and will also be counted as non-responder (Not Evaluable for Response), instead of counted as missing.

# Criteria for Evaluation: **Efficacy measurements**:

 ORR is defined as the percentage of subjects who have achieved confirmed CR and PR during treatment phase, according to RECIST v1.1. Not-confirmed CR or PR, or withdraw for DLT are counted as non-responder.

#### 2 Mock-up Tables and Figures

The Mock-up "TABLES and FIGURES" is planned according to ICH E3, in which relevant CSR section is 14. The words shadowed below are to be adjusted or repeated upon real data, or just for notification.

For all statistical analyses tables, the descriptive statistics will be displayed on maximum treatment dose level and overall.

Columns {Label, Max. Dose Levels, Total} will be included with the analyzed population specified. In the mock table below, only the Label with one treatment column were presented to show the descriptive/inferential statistics to be displayed in the final tabulation.



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

The DSMB, composed of medical monitors (physicians experienced in oncology studies) and at least one statistician. Their responsibilities are to review and evaluate the data for safety, study conduct and progress, and make recommendations concerning the continuation, modification, or termination of study. Serial assessments of PK results also may be taken into account for safety evaluation. A neurologist will be invited to join DSMB meeting as a consultant when neurotoxicity occurred.

The document review or meeting of DSMB will be held when the following scenarios:

- A subject is not recovered from Grade 2 neurotoxicity over three weeks;
- A subject revealed Grade 3 or above neurotoxicity;
- After 10 evaluable subjects finished the study in Stage I

#### Note:

(1) Site ID:

| Site ID | Site Name |
|---------|-------------------------------------------------------|
| 1 | Taipei Medical University Hospital (TMUH) |
| 2 | National Cheng Kung University Hospital (NCKUH) |
| 3 | Taipei Veterans General Hospital (TVGH) |
| 4 | Taipei Medical University Shuang Ho Hospital (TMUSHH) |

- (2) Study subjects will be categorized into the following populations for analysis:
  - Intention-to-treat (ITT) population: The ITT population consists of all subjects enrolled in the study and received at least one study treatment.
  - Per-protocol (PP) population: The PP population will consist of all subjects who
    - (1) withdraw from study for DLT, or
    - (2) completed at least 3 cycles of study treatment regimen, have measurable baseline disease and, at least, one post-baseline RECIST assessment (PD, SD, PR or CR). Subjects with a major protocol deviation or AE, deemed by the Medical Monitor to have an impact on the study endpoints, will be excluded from the PP population.
  - PK population: The PK population will consist of all subjects in stage I who received, at least, one dose of 24 mg/m<sup>2</sup> of SCB01A with sufficient post-dose bio-samples collected for PK profile characterization.
- (3) Maximum treatment dose level

Level 1 (12 mg/m²) Level 1a (9 mg/m²) Level 1b (7 mg/m²) Level 2 (18 mg/m²) Level 2a (15 mg/m²) Level 2b (12 mg/m²) Level 3 (24 mg/m²) Level 3a (20 mg/m²) Level 3b (16 mg/m²)

(4) For Visit Name, C(c) denotes cycle (c), D(d) denotes day (d)

| ` | Visit Name, C(c) denotes eyele (c), B(d) denotes day (d) | | |
|---|---|---|---|
| Visit No. | Visit Name | Code | Planned Visit Day |
| 0 | Screening Visit | SV | <b>-28</b> ∼ <b>-1</b> |
| 1.01 | Cycle 1 Day 1 | C1D1 | 1 |
| 1.08 | Cycle 1 Day 8 | C1D8 | 7±1 days after C1D1 |
| 1.15 | Cycle 1 Day 15 | C1D15 | 14±2 days after C1D1 |
| c.01 | Cycle © Day 1 | CcD1 | 21±1 days after Ck1D1<br>k=c-1 |
| c.08 | Cycle © Day 8 | CcD8 | 7±1 days after CcD1 |
| c.15 | Cycle © Day 15, ©=1, 2, 3 only | CcD15 | 14±2 days after CcD1 |
| | End of Treatment (EOT) / Early Withdrawal (EW) | EOT /<br>EW | EOT: 21±2 days after Ck1D1 or 14±2 days after Ck1D8, k=c-1 EW: after the last treatment dose |
| 99.1 | Follow-Up Visit 1 (FU1) | FU1 | 21±3 after EOT/EW |
| 99.2 | Follow-Up Visit 2 (FU2) | FU2 | 21±3 after FU1-W3 |

Version 3.0, 14DEC2018 Protocol No.: SCB01A-22 

SynCore Biotechnology Co., Ltd. Prepared by: A2 Healthcare Taiwan Corporation



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Visit No. | Visit Name | Visit<br>Code | Planned Visit Day |
|-----------|-------------------------|---------------|-----------------------|
| 99.3 | Follow-Up Visit 3 (FU3) | FU3 | 21±3 after FU2-W6 |
| 99. F | Follow-Up Visit F (FUF) | FU[F] | Every 9 weeks ±7 days |
| 66.XX | Unscheduled Visit (UV) | UV | |

 $<sup>\</sup>boxed{c}$ : cycle number where  $\boxed{c} \ge 2$ ,  $\boxed{F}$ : assigned sequentially from 4,  $\boxed{x}$ : assigned sequentially from 01

(5) Full term for 'Protocol Deviation Code':

| Code | Full Term |
|------|-------------------------------------------------|
| | To be added upon real data in final tabulation> |

(6) Clinical description of severity for CTCAE Term:

| CTCAE Term | Clinical description |
|------------------------------|-----------------------------------|
| Tachycardia | Heart rate > 100 bpm |
| Bradycardia | Heart rate < 60 bpm |
| Hypertension Grade ≥1 | SBP > 120 or DBP > 80 mmHg |
| Hypertension Grade ≥2 | SBP > 140 or DBP > 90 mmHg |
| Hypertension Grade ≥3 | SBP > 160 or DBP > 100 mmHg |
| Hypotension | SBP < 90 or DBP < 60 mmHg |
| Fever Grade ≥1 | Temperature $\geq$ 38 degree C |
| Fever Grade ≥3 | Temperature $\geq 40$ degree C |
| Hypothermia Grade ≥2 | temperature ≤ 35 degree C |
| Hypothermia Grade ≥3 | temperature ≤ 32 degree C |
| Tachypnea | respiratory rate > 20 breaths/min |
| Bradypnea | respiratory rate < 12 breaths/min |
| QTc Prolonged Grade ≥ 1 | $QTc \ge 450 \text{ msec}$ |
| QTc Prolonged Grade $\geq 3$ | $QTc \ge 501 \text{ msec}$ |

(7) For clinical relevant

CS: abnormal and clinically significant LLN: lower limit of normal range NCS: abnormal but not clinically significant ULN: upper limit of normal range

(8) Abbreviations of statistics

N: number of non-missing values

ANOVA: analysis of variance

ANCOVA: analysis of covariance

Mean: mean of values CHISQ: Chi-Square test

SD: standard deviation of values CMH: Cochran-Mantel-Haenszel test adjusted by stratification

Q1: 25% quartile of values

CMH[G]: CMH for General Association

CMH[D]: CMH for Row Mean Scores Differ

Median: median of values FISHER: Fisher's exact test IQR: inter-quartile-range (IQR=Q3-Q1) KW: Kruskal-Wallis test

Min: minimum of values MHCHISQ: Mantel-Haenszel chi-square test on given scores

Max: maximum of values T: two sample t test

CI: confidence interval W: Wilcoxon Rank-sum Test

LS-mean: least-square mean Diff.: difference

#### 3 Change From Preceding Version of Statistical Analysis Plan

#### 3.1 SAP 2.0: Progression Free Survival (PFS) Estimation

For Progression Free Survival, missing data will be estimated as the time from treatment onset date to date of last implementation of radiological image assessment +1 or estimated as '1' if no post-treatment tumor assessment available. Estimating missing data as censored on Day 1 shall be rather conservative than omitting the missing ones.

### 

# Statistical Analysis Plan: Mock-up Tables and Figures

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### 6.1. Efficacy Measurements

Subjects will be considered evaluable for tumor assessment in this study if they fulfill the criteria for evaluation according to RECIST v1.1, i.e., those subjects who undergo a baseline disease assessment within 4 weeks of treatment initiation, and who undergo at least 1 disease assessment on study (the following should be revised if revision in corresponding part in synopsis is accepted).

• PFS is defined as the time from the start of treatment up to the date of first progression based on RECIST v1.1 or the date of death, whichever comes first.

#### 3.2 SAP 3.0: Response Evaluation

There are 5 subjects who are not evaluated due to clinical disease progression or AE/SAE. The subjects will be counted as 'Not Evaluable for Response' if no any post-treatment radiological image assessments. Each patient will be assigned one of the following categories:

- 1. Complete response
- 2. Partial response
- 3. Stable disease
- 4. Progression disease
- 5. Not Evaluable for Response.



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### 14 TABLES AND FIGURES

#### 14.1 DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS

#### 14.1.1 Screen Failures and Subject Disposition by Study Site

| Characteristics | Study Site |
|--------------------------------------------|-------------|
| All Screened Subjects (multiple-selection) | |
| N | XXX |
| Eligible Subjects | XXX (XXX.X% |
| Screening Failures | XXX (XXX.X% |
| ~INC01 | XXX (XXX.X% |
| ~INC02 | XXX (XXX.X% |
| ~INC03 | XXX (XXX.X% |
| ~EXC01 | XXX (XXX.X% |
| ~EXC02 | XXX (XXX.X% |
| ~EXC03 | XXX (XXX.X% |
| Eligible Subject (multiple-selection) | |
| N | XXX |
| ~ ITT | XXX (XXX.X% |
| ~ PP | XXX (XXX.X% |
| ~ Non-PP | XXX (XXX.X% |
| ~ < Reason 1> | XXX (XXX.X% |
| ~ < Reason 2> | XXX (XXX.X% |
| | XXX (XXX.X% |
| ~ Non-ITT | XXX (XXX.X% |

# 14.1.2 Study Visits, Study Termination, Subject Disposition and Protocol Deviation

Population: ITT Population

| Characteristics | Max. Dose Level |
|-----------------------------------------------|-----------------|
| . Study Termination | |
| N | XXX |
| Study Completed | XXX (XXX.X%) |
| Prematurely Discontinued | XXX (XXX.X%) |
| ~ Withdrew consent | XXX (XXX.X%) |
| $\sim$ AE | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| . Study visits completed (multiple-selection) | |
| N | XXX |
| Screening Visit (SV) | XXX (XXX.X%) |
| Cycle 1 Day 1 (C1D1) | XXX (XXX.X%) |
| Cycle 1 Day 8 (C1D8) | XXX (XXX.X%) |
| Cycle 1 Day 15 (C1D15) | XXX (XXX.X%) |
| Cycle © Day 1 (C©D1) | XXX (XXX.X%) |
| Cycle © Day 8 (C©D8) | XXX (XXX.X%) |
| Cycle © Day 15 (C©D15) | XXX (XXX.X%) |
| End of Treatment (EOT) /Early Withdrawal (EW) | XXX (XXX.X%) |
| Toxicity Follow-Up Visit (TFU) | XXX (XXX.X%) |



# **Statistical Analysis Plan: Mock-up Tables and Figures** SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|------------------------------------------|-----------------|
| . Study Duration [days] | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| .Population (multiple-selection) | |
| N | XXX |
| ~ PP | XXX (XXX.X%) |
| ~ Non-PP | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| .Protocol Deviation (multiple-selection) | |
| N | XXX |
| ~ Major Protocol Deviation | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| ~ Minor Protocol Deviation | XXX (XXX.X%) |
| ~ < Reason 1> | XXX (XXX.X%) |
| ~ < Reason 2> | XXX (XXX.X%) |
| | XXX (XXX.X%) |

Study Duration [days] = End Date of Treatment Phase - Visit 0, or alternatively as the last visit date - Visit 0

#### 14.1.3 Demographic Data, Smoking Status and Betelnut Consumption

| Characteristics | Max. Dose Level |
|--------------------------------------------------|------------------------|
| Study Site | |
| N | XXX |
| Site 01: TMUH | XXX (XXX.X%) |
| Site 02: NCKUH | XXX (XXX.X%) |
| Site 03: TVGH | XXX (XXX.X%) |
| Site 04: TMUSHH | XXX (XXX.X%) |
| . Variable, including Age [Y/O], Body Weight [kg | g], Body Height [cm], |
| BMI [kg/m^2]<br>N (Missing) | VVV (VVV) |
| Mean (SD) | XXX (XXX)<br>XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| . Gender | |
| N (Missing) | XXX (XXX) |
| Male | XXX (XXX.X%) |
| Female | XXX (XXX.X%) |
| . Race | |
| N (Missing) | XXX (XXX) |

SynCore Biotechnology Co., Ltd. Version 3.0, 14DEC2018 Confidential Prepared by: A2 Healthcare Taiwan Corporation Protocol No.: SCB01A-22 



# **Statistical Analysis Plan:** Mock-up Tables and Figures SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|--------------------------|-----------------|
| Aboriginal | XXX (XXX.X%) |
| Asian | XXX (XXX.X%) |
| Black / African American | XXX (XXX.X%) |
| Torres Strait Islander | XXX (XXX.X%) |
| White or Caucasian | XXX (XXX.X%) |
| Other | XXX (XXX.X%) |
| . Ethnicity | |
| N (Missing) | XXX (XXX) |
| Hispanic or Latino | XXX (XXX.X%) |
| Not Hispanic/Latino | XXX (XXX.X%) |
| . Smoking Status | |
| N (Missing) | XXX (XXX) |
| Never Smoked | XXX (XXX.X%) |
| Former Smoker | XXX (XXX.X%) |
| Current Smoker | XXX (XXX.X%) |
| . Betelnut Consumption | |
| N (Missing) | XXX (XXX) |
| Never Took Betelnut | XXX (XXX.X%) |
| Former Taker | XXX (XXX.X%) |
| Current Taker | XXX (XXX.X%) |

Age [Y/O] = year of informed consent – year of birth BMI  $[kg/m^2]$  = Body Weight  $[kg]/(Body Height [cm]/100)^2$ 

#### 14.1.4 Head and Neck Squamous Cell Carcinoma History & Tumor **Staging**

| Staging | |
|-----------------------------------------|-----------------|
| Population: ITT Population | |
| Characteristics | Max. Dose Level |
| . Disease Duration [Years] | |
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | $XXX\sim XXX$ |
| Min~Max | XXX~XXX |
| . Disease Status (multiple-selection) | |
| N (Missing) | XXX (XXX) |
| Recurrence | XXX (XXX.X%) |
| Disease Progression | XXX (XXX.X%) |
| Metastasis | XXX (XXX.X%) |
| . Histological grade | |
| N (Missing) | XXX (XXX) |
| Cannot be assessed | XXX (XXX.X%) |
| Undifferentiated | XXX (XXX.X%) |
| Poorly differentiated | XXX (XXX.X%) |
| Moderate differentiated | XXX (XXX.X%) |
| Well differentiated | XXX (XXX.X%) |
| . Metastatic sites (multiple-selection) | |
| N (Missing) | XXX (XXX) |

SynCore Biotechnology Co., Ltd. Version 3.0, 14DEC2018 Confidential Prepared by: A2 Healthcare Taiwan Corporation Protocol No.: SCB01A-22 



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|-----------------|-----------------|
| Lymph | XXX (XXX.X%) |
| Mediastinum | XXX (XXX.X%) |
| Bone | XXX (XXX.X%) |
| Bone Marrow | XXX (XXX.X%) |
| Adrenal | XXX (XXX.X%) |
| Nodes Lung | XXX (XXX.X%) |
| Liver | XXX (XXX.X%) |
| Skin | XXX (XXX.X%) |
| Chest Wall | XXX (XXX.X%) |
| CNS | XXX (XXX.X%) |
| Other | XXX (XXX.X%) |
| . Tumor Stage | |
| N (Missing) | XXX (XXX) |
| Stage I | XXX (XXX.X%) |
| Stage II | XXX (XXX.X%) |
| Stage III | XXX (XXX.X%) |
| Stage IVa | XXX (XXX.X%) |
| Stage IVb | XXX (XXX.X%) |

Disease Duration [years] = (date of screening visit – earliest onset date of initial diagnosis with histological or cytological confirmation)/365.25, missing day is estimated as 15, missing month is estimated as Jul-01

#### 14.1.5 General Medical History

| Characteristics | Max. Dose Level |
|-----------------------------------------|-----------------|
| .Medical History (multiple-selection) | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| ~ Ophthalmologic | XXX (XXX.X%) |
| ~ Ear, Nose, Throat, Mouth | XXX (XXX.X%) |
| ~ Cardiovascular | XXX (XXX.X%) |
| ~ Cerebrovascular | XXX (XXX.X%) |
| .Current Condition (multiple-selection) | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| ~ Ophthalmologic | XXX (XXX.X%) |
| ~ Ear, Nose, Throat, Mouth | XXX (XXX.X%) |
| ~ Cardiovascular | XXX (XXX.X%) |
| ~ Cerebrovascular | XXX (XXX.X%) |

Current condition lists the medical histories that are ongoing or with end date  $\geq$  date of visit 0

#### 14.1.6 Study Drug Administration

Population: ITT Population

Characteristics Max. Dose Level

Maximum Unit Dose Level [mg/m^2], Maximum Unit Dose [mg],

Cumulated Dose Level [mg/m^2], Cumulated Dose [mg],

 $Mean\ Cycle\ Dose\ Level\ [mg/m^2/cycle],\ Mean\ Cycle\ Dose\ [mg/cycle]$ 

<sup>.</sup> Treatment Exposure [cycles],



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|-----------------|-----------------|
| N (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | $XXX\sim XXX$ |
| Min~Max | XXX~XXX |

For Treatment Exposure, completion of Day 1 and Day 8 is counted as 1 cycle, and Day 1 only is counted as 0.5 cycle.

#### 14.2 EFFICACY DATA

By stage analysis, no Overall of both stages will be presented if only stage I data are available.

#### 14.2.1 Objective Response Rate

| opulation: ITT / PP Population | |
|----------------------------------------------------------|-----------------|
| Characteristics | Max. Dose Level |
| Stage: Overall, Stage I, Stage II | |
| Population: ITT, PP | |
| Best Response | |
| N (Missing) | XXX (XXX) |
| CR | XXX (XXX.X%) |
| PR | XXX (XXX.X%) |
| ORR(CR + PR) | XXX (XXX.X%) |
| SD | XXX (XXX.X%) |
| PD | XXX (XXX.X%) |
| Not Evaluable for Response | XXX (XXX.X%) |
| 95% CI of ORR (WI) | XXX-XXXb |
| . Any PD for Target Lesions | |
| . Any PD for Non-Target Lesions | |
| . Any PD for Overall Response | |
| N (Missing) | XXX (XXX) |
| Yes | XXX (XXX.X%) |
| No | XXX (XXX.X%) |
| Progression Free Survival [days], Overall Survival[days] | |
| N (Missing) | XXX (XXX) |
| Censored No. | XXX (XXX%) |
| Observed No. | XXX (XXX%) |
| Q1 [95% CI] | XXX [XX~XX] |
| Median [95% CI] | XXX [XX~XX] |
| Q3 [95% CI] | XXX XX~XX |

For CI (WI, within group), b denotes exact CI of binomial proportion of # using binomial test Progression Free Survival [days] = Date of PD / death – treatment onset date + 1, or date of Last Implementation of Radiological Image Assessment – treatment onset date + 1, or estimated as '1' if no post-treatment tumor assessment available.

Overall Survival[days] = Date of death – treatment onset date +1, or last known alive date – treatment onset date +1

#### 14.2.1.1 Kaplan-Meier Graph on Progression Free Survival (ITT)

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### 14.2.1.2 Kaplan-Meier Graph on Progression Free Survival (PP)

#### 14.2.1.3 Kaplan-Meier Graph on Overall Survival (ITT)





#### 14.3 SAFETY DATA

#### 14.3.1 Treatment Emergent Adverse Events – Subject Based Analyses

#### 14.3.1.1 Treatment Emergent AEs – Subjects with AEs

#### 14.3.1.2 Treatment Emergent AEs – Subjects with DLTs

Population: ITT Population Characteristics Max. Dose Level . By MedDRA SOC and Preferred Term XXXAt least one below XXX (XXX.X%) <MedDRA Body System1> XXX (XXX.X%) ~ < MedDRA Preferred Term 1> XXX (XXX.X%) ~ < MedDRA Preferred Term 2> XXX (XXX.X%) ~ < MedDRA Preferred Term 3> XXX (XXX.X%) <MedDRA Body System2> XXX (XXX.X%) ~ < MedDRA Preferred Term 1> XXX (XXX.X%) ~ < MedDRA Preferred Term 2> XXX (XXX.X%) ~ < MedDRA Preferred Term 3> XXX (XXX.X%)

#### For each MedDRA SOC or Preferred Term, Subject with multiple events are counted as one incidence.

#### 14.3.1.3 Treatment Emergent AEs – Subjects with Grade ≥3 AEs

Population: ITT Population

| <u> </u> | |
|------------------------------------|-----------------|
| Characteristics | Max. Dose Level |
| . By MedDRA SOC and Preferred Term | |
| N | XXX |



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|--------------------------------------|-----------------|
| At least one below | XXX (XXX.X%) |
| <meddra body="" system1=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| $Grade \ge 4$ | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX (XXX.X%) |
| $Grade \ge 4$ | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX (XXX.X%) |
| <meddra body="" system2=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX (XXX.X%) |

#### Grade $\geq$ 4 AEs will be listed additionally if any

#### 14.3.1.4 Treatment Emergent AEs – Subject with Treatment Related AEs

Population: ITT Population

| Characteristics | Max. Dose Level |
|--------------------------------------|-----------------|
| . By MedDRA SOC and Preferred Term | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| <meddra body="" system1=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX (XXX.X%) |
| <meddra body="" system2=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX (XXX.X%) |

Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related

#### 14.3.1.5 Treatment Emergent AEs – Subject with Treatment Modified AEs

Population: ITT Population

| Characteristics | Max. Dose Level |
|---------------------------------------------------|-----------------|
| The Action Taken by MedDRA SOC and Preferred Term | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| <meddra body="" system1=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ Treatment Infusion Interrupted | XXX (XXX.X%) |
| ~ Treatment Omitted | XXX (XXX.X%) |
| ~ Dose Reduced | XXX (XXX.X%) |
| ~ Treatment Discontinued | XXX (XXX.X%) |
| <meddra body="" system2=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ Treatment Infusion Interrupted | XXX (XXX.X%) |
| ~ Treatment Omitted | XXX (XXX.X%) |
| ~ Dose Reduced | XXX (XXX.X%) |
| ~ Treatment Discontinued | XXX (XXX.X%) |



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### 14.3.1.6 Treatment Emergent AEs – Subjects with SAEs

Population: ITT Population

| Characteristics | Max. Dose Level |
|----------------------------------------|-----------------|
| . By MedDRA SOC and Preferred Term | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| <meddra body="" system1=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX (XXX.X%) |
| ~ Death | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX (XXX.X%) |
| ~ Death | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX (XXX.X%) |
| ~ Death | XXX (XXX.X%) |
| <meddra body="" system2=""></meddra> | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 1> | XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX (XXX.X%) |
| ~ Death | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 2> | XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX (XXX.X%) |
| ~ Death | XXX (XXX.X%) |
| ~ < MedDRA Preferred Term 3> | XXX (XXX.X%) |
| ~ Requires or Prolongs Hospitalization | XXX (XXX.X%) |
| ~ Death | XXX (XXX.X%) |

# SynCoreBio

#### Statistical Analysis Plan: Mock-up Tables and Figures

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| 14.3.2 Clinical Relevance of Laboratory | Assessment – Hematology |
|-----------------------------------------|-------------------------|
|-----------------------------------------|-------------------------|

- 14.3.2.1 Clinical Relevance of Hematology Item 1
- 14.3.2.2 Clinical Relevance of Hematology Item 2
- 14.3.2.3 ...

#### 14.3.3 Clinical Relevance of Laboratory Assessment – Biochemistry

- 14.3.3.1 Clinical Relevance of Biochemistry Item 1
- 14.3.3.2 Clinical Relevance of Biochemistry Item 2
- 14.3.3.3 ...

#### 14.3.4 Clinical Relevance of Laboratory Assessment – Coagulation

- 14.3.4.1 Clinical Relevance of Coagulation Item 1
- 14.3.4.2 Clinical Relevance of Coagulation Item 2
- 14.3.4.3 ...

#### 14.3.5 Clinical Relevance of Laboratory Assessment – Urinalysis

- 14.3.5.1 Clinical Relevance of Urinalysis Item 1
- 14.3.5.2 Clinical Relevance of Urinalysis Item 2
- 14.3.5.3 ...

Population: ITT Population

Characteristics

| Characteristics | Wax. Dose Level |
|---------------------------------------------------|------------------------|
| The Warst Clinical Paleyanes of Pagaline Labor | otom |
| The Worst Clinical Relevance of Baseline Labor | |
| (Baseline visits are Screening Visit, Cycle 1 Day | · |
| N | XXX |
| Normal | XXX (XXX.X%) |
| NCS | XXX (XXX.X%) |
| CS | XXX (XXX.X%) |
| The Worst Clinical Relevance of Post-Baseline I | Laboratory |
| (Excluding Baseline Visits) | Ž |
| N | XXX |
| Normal | XXX (XXX.X%) |
| NCS | XXX (XXX.X%) |
| CS | XXX (XXX.X%) |
| The Worst Clinical Relevance Change from Base | eline to Post-Baseline |
| N (Missing) | XXX (XXX) |
| Relieved: CS to Normal / NCS | XXX (XXX.X%) |
| Unchanged | XXX (XXX.X%) |
| Worsened: Normal / NCS to CS | XXX (XXX.X%) |

Max Dose Level

Unchanged: Normal to Normal, NCS to NCS, Normal to NCS, NCS to Normal

Baseline visits are Screening Visit, Cycle 1 Day 1

The Worst Clinical Relevance of Baseline : Compare the data in the two Baseline visits and list the worst one Worst: CS > NCS > Normal

#### 14.3.6 Toxicity Grade of Laboratory Assessment – Hematology



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| 14.3.6.1 | Toxicity Grade of Hematology – Item 1 | |
|---|---|---|
| 14.3.6.2 | Toxicity Grade of Hematology – Item 2 | |
| 14.3.6.3 | ••• | |
| .3.7 Toxic | ity Grade of Laboratory Assessmen | t – Biochemistry |
| 14.3.7.1 | Toxicity Grade of Biochemistry – Item 1 | • |
| 14.3.7.2 | Toxicity Grade of Biochemistry – Item 2 | |
| 14.3.7.3 | · | |
| I.3.8 Toxici | ty Grade of Laboratory Assessmen | t – Coagulation |
| 14.3.8.1 | Toxicity Grade of Coagulation – Item 1 | |
| 14.3.8.2 | Toxicity Grade of Coagulation – Item 2 | |
| 14.3.8.3 | ••• | |
| 4.3.9 Toxici | ity Grade of Laboratory Assessmen | t –Urinalysis |
| 14.3.9.1 | Toxicity Grade of Urinalysis – Item 1 | · |
| 14.3.9.2 | Toxicity Grade of Urinalysis – Item 2 | |
| 14.3.9.3 | | |
| opulation: ITT<br>Characteristics | Population | Max. Dose Level |
| The Worst Tox | icity Grade of Baseline Laboratory | |
| | are Screening Visit, Cycle 1 Day 1) | |
| N | | XXX |
| Grade 0 | | XXX (XXX.X%) |
| Grade 1<br>Grade 2 | | XXX (XXX.X%)<br>XXX (XXX.X%) |
| Grade 3 | | XXX (XXX.X%) |
| The Worst Tox | icity Grade of Post-Baseline Laboratory | |
| (Excluding Bas | eline Visits) | |
| N | | XXX |
| Grade 0 | | XXX (XXX.X%) |
| Grade 1 | | XXX (XXX.X%) |
| Grade 2 | | XXX (XXX.X%) |
| Grade 3 | | XXX (XXX.X%) |
| ••• | | ••• |
| The Worst Tox | icity Grade Change: Post-Baseline - Baseline | |
| N | | XXX |
| Grade +3 | | XXX (XXX.X%) |
| Consider 12 | | |

Visits with Toxicity Grade Change ≥ Grade +3

Grade +2

Grade +1

Grade 0

Grade -1

Grade -2

Version 3.0, 14DEC2018 Confidential SynCore Biotechnology Co., Ltd. Prepared by: A2 Healthcare Taiwan Corporation

XXX (XXX.X%)

XXX (XXX.X%)

XXX (XXX.X%)

XXX (XXX.X%)

XXX (XXX.X%)



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|-----------------|-----------------|
| N | XXX |
| Cycle 1 Day 1 | XXX (XXX.X%) |
| Cycle 1 Day 8 | XXX (XXX.X%) |
| Cycle 1 Day 15 | XXX (XXX.X%) |
| ••• | ••• |

Baseline visits are Screening Visit, Cycle 1 Day 1

The Worst Clinical Relevance of Baseline: Compare the data in the two Baseline visits and list the worst one Worst: Grade 5 > Grade 4 > Grade 3 > Grade 2 > Grade 1 > Grade 0

#### 14.3.10 Vital Signs, Body Weight and ECOG Performance Status

| 14.3.10.1 | Heart Rate [bpr | nl |
|-----------|-----------------|----|
| 14.5.10.1 | neart Kate iddi | ш |

14.3.10.2 Systolic Blood Pressure and Diastolic Blood Pressure [mmHg]

14.3.10.3 Temperature [Degree C]

14.3.10.4 Respiratory Rate [breaths/min]

14.3.10.5 Weight [kg]

| Population: | ΙT | ΤP | opu | lation |
|-------------|----|----|-----|--------|
|-------------|----|----|-----|--------|

(Excluding Baseline Visits)

| Max. Dose Level |
|---|
| s Screening |
| XXX |
| XXX (XXX) |
| XXX (XXX) |
| XXX~XXX |
| XXX~XXX |
| on) |
| as |
| and the second s |
| XXX |
| XXX (XXX.X%) |
| 71111 (11111.1170) |
| XXX (XXX.X%) |
| · |
| XXX (XXX.X%) |

Version 3.0, 14DEC2018 Confidential SynCore Biotechnology Co., Ltd. Prepared by: A2 Healthcare Taiwan Corporation

XXX



Mock-up Tables and Figures
SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|---|---|
| At least one below | XXX (XXX.X%) |
| Tachycardia | XXX (XXX.X%) |
| Bradycardia | XXX (XXX.X%) |
| Hypertension Grade $\geq 1$ | XXX (XXX.X%) |
| Hypertension Grade $\geq 2$ | XXX (XXX.X%) |
| Hypertension Grade $\geq 3$ | XXX (XXX.X%) |
| Hypotension | XXX (XXX.X%) |
| Fever Grade ≥1 | XXX (XXX.X%) |
| Fever Grade ≥3 | XXX (XXX.X%) |
| Hypothermia Grade ≥2 | XXX (XXX.X%) |
| Hypothermia Grade ≥3 | XXX (XXX.X%) |
| Tachypnea | XXX (XXX.X%) |
| Bradypnea | , |
| Vital Signs Significant Change from Baseline to Post-Baseline Visi | ts |
| (multiple-selection) | |
| N | XXX |
| At least one below | XXX (XXX.X%) |
| Non-Tachycardia to Tachycardia | XXX (XXX.X%) |
| ~ Cycle 1 Day 1 | XXX (XXX.X%) |
| ~ Cycle 1 Day 8 | XXX (XXX.X%) |
| ~ Cycle 1 Day 15 | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| Non-Bradycardia to Bradycardia | |
| Non-Hypertension Grade $\leq 2$ to Hypertension Grade $\geq 2$ | |
| Hypertension Grade $\leq 3$ to Hypertension Grade $\geq 3$ | |
| Non-Hypotension to Hypotension | |
| Non-Fever Grade=0 to Fever Grade ≥1 | |
| Non-Fever Grade $\leq 3$ to Fever Grade $\geq 3$ | |
| Non-Hypothermia Grade<2 to Hypothermia Grade≥2 | |
| Non-Hypothermia Grade<3 to Hypothermia Grade≥3<br>Non-Tachypnea to Tachypnea | |
| Non-1acnypnea to 1acnypnea<br>Non-Bradypnea to Bradypnea | |
| Non-Bradypnea to Bradypnea The same layout as above> | |
| Resoline is Cycle 1 Day 1 (Pre IV Infusion) or alternatively as Screen | ming Vigit if Cycle 1 Day 1 data is not |

Baseline is Cycle 1 Day 1 (Pre-IV Infusion) or alternatively as Screening Visit if Cycle 1 Day 1 data is not available.

#### 14.3.10.6 ECOG Performance Status

| Population: ITT Population | |
|---|---|
| Characteristics | Max. Dose Level |
| The Worst ECOG Performance Status at Baseline Vis | its (multiple- |
| selection) | |
| (Baseline visits are Screening Visit, Cycle 1 Day 1) | |
| N | XXX |
| ECOG≥1 | XXX (XXX.X%) |
| ECOG ≥2 | XXX (XXX.X%) |
| ECOG≥3 | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| The Worst ECOG Performance Status at Post-Baselin selection) (Excluding Baseline Visits) | e Visits (multiple- |
| N | XXX |

Version 3.0, 14DEC2018 Confidential SynCore Biotechnology Co., Ltd. Protocol No.: SCB01A-22  Prepared by: A2 Healthcare Taiwan Corporation



SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|-----------------------------------------------|---------------------|
| ECOG ≥1 | XXX (XXX.X%) |
| ECOG ≥2 | XXX (XXX.X%) |
| ECOG≥3 | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| The Worst ECOG Performance Status Change from | n Baseline to Post- |
| Baseline Visits (multiple-selection) | |
| N | XXX |
| At least one below | XXX |
| ECOG <1 to ECOG ≥1 | XXX (XXX.X%) |
| Cycle 1 Day 1 | XXX (XXX.X%) |
| Cycle 1 Day 8 | XXX (XXX.X%) |
| Cycle 1 Day 15 | XXX (XXX.X%) |
| ECOG <2 to ECOG ≥2 | XXX (XXX.X%) |
| Cycle 1 Day 1 | XXX (XXX.X%) |
| Cycle 1 Day 8 | XXX (XXX.X%) |
| Cycle 1 Day 15 | XXX (XXX.X%) |

Baseline visits are Screening Visit, Cycle 1 Day 1

The Worst Clinical Relevance of Baseline: Compare the data in the two Baseline visits and list the worst one Worst: Grade 5 > Grade 4 > Grade 3 > Grade 2 > Grade 1 > Grade 0

#### 14.3.11 Nerve Conduction Velocity Examination

- 14.3.11.1 Neurosensory Result
- 14.3.11.2 Neuromotor Result

<Use the layout for 14.3.2 Clinical Relevance of Laboratory Assessment – Hematology>

#### 14.3.12 Electrocardiogram (ECG, EKG)

#### 14.3.12.1 Electrocardiogram - Overall Interpretation

<Use the layout for 14.3.2 Clinical Relevance of Laboratory Assessment – Hematology>

- 14.3.12.2 Electrocardiogram PR Interval [msec]
- 14.3.12.3 Electrocardiogram QRS Interval [msec]

#### 14.3.12.4 Electrocardiogram - QTc Interval [msec]

Population: ITT Population

| 1 opulation: 11 1 opulation | |
|---|---|
| Characteristics | Max. Dose Level |
| Baseline Value | |
| (Baseline is Cycle 1 Day 1 (Pre-IV Infusion) or alternatively as | |
| Screening Visit if Cycle 1 Day 1 data is not available) | |
| N | XXX |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | $XXX\sim XXX$ |
| Min~Max | XXX~XXX |

ECG Abnormalities at Baseline Visits (multiple-selection) (Baseline is Cycle 1 Day 1 (Pre-IV Infusion) or alternatively as Screening Visit if Cycle 1 Day 1 data is not available)



**Mock-up Tables and Figures** SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|---|---|
| N | XXX |
| QTc Prolonged Grade $\geq 1$ | XXX (XXX.X%) |
| QTc Prolonged Grade $\geq 3$ | XXX (XXX.X%) |
| ECG Abnormalities at Post-Baseline Visits (multiple-selection) | |
| (Excluding Baseline Visits) | |
| N | XXX |
| QTc Prolonged Grade $\geq 1$ | XXX (XXX.X%) |
| QTc Prolonged Grade $\geq 3$ | XXX (XXX.X%) |
| ECG Significant Change from Baseline to Post-Baseline Visits (multiple- | |
| selection) | 3/3/3/ |
| N | XXX |
| At least one below | XXX |
| QTc Prolonged Grade $\leq 1$ to Grade $\geq 1$ | XXX (XXX.X%) |
| ~ Cycle 1 Day 1 | XXX (XXX.X%) |
| ~ Cycle 1 Day 8 | XXX (XXX.X%) |
| ~ Cycle 1 Day 15 | XXX (XXX.X%) |
| QTc Prolonged Grade $\leq 3$ to Grade $\geq 3$ | XXX (XXX.X%) |
| ~ Cycle 1 Day 1 | XXX (XXX.X%) |
| ~ Cycle 1 Day 8 | XXX (XXX.X%) |
| ~ Cycle 1 Day 15 | XXX (XXX.X%) |

Baseline is Cycle 1 Day 1 (Pre-IV Infusion) or alternatively as Screening Visit if Cycle 1 Day 1 data is not available.

#### 14.3.13 Physical Examination

# 14.3.13.1 Physical Examination – All Abnormalities Population: ITT Population

| Characteristics | Max. Dose Level |
|-----------------------------------------------------|-----------------|
| The Worst Physical Abnormalities at Baseline | |
| Baseline visits are Screening Visit, Cycle 1 Day 1) | |
| N (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| The Worst Physical Abnormalities at Post-Basel | ine |
| Excluding Baseline Visits) | |
| N (Missing) | XXX(XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| ••• | XXX (XXX.X%) |



### **Statistical Analysis Plan:** Mock-up Tables and Figures SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Characteristics | Max. Dose Level |
|---|---|
| ransition of the Worst Physical Abnormalities from Baseline to Post-Baseline (Normal to NCs | |
| CS) | |
| N (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| | XXX (XXX.X%) |

The Worst Clinical Relevance of Baseline: Compare the data in the two Baseline visits and list the worst one Worst: CS > NCS > Normal

#### Physical Examination - Clinical Significant (CS) Abnormalities 14.3.13.2

Population: ITT Population

| Characteristics | Max. Dose Level |
|------------------------------------------------------|-----------------|
| The Worst CS Physical Abnormalities at Baselin | ne |
| (Baseline visits are Screening Visit, Cycle 1 Day 1) | |
| N (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| The Worst CS Physical Abnormalities at Post-B | aseline |
| (Excluding Baseline Visits) | |
| N (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| | XXX (XXX.X%) |

#### Transition of the Worst CS Physical Abnormalities from Baseline to Post-Baseline (Normal/NCS to CS)

| N (Missing) | XXX (XXX) |
|--------------------------------|--------------|
| At least one below | XXX (XXX.X%) |
| ~ <body 1="" system=""></body> | XXX (XXX.X%) |
| ~ <body 2="" system=""></body> | XXX (XXX.X%) |
| ~ <body 3="" system=""></body> | XXX (XXX.X%) |
| ~ <body 4="" system=""></body> | XXX (XXX.X%) |
| | XXX (XXX.X%) |

The Worst Clinical Relevance of Baseline: Compare the data in the two Baseline visits and list the worst one Worst: CS > NCS > Normal